CLINICAL TRIAL: NCT01099982
Title: Assessing Changes in Myocardial Tissue and Blood in Patients With Advanced Heart Disease, Effects of Mechanical Unloading on Myocardial Function and Structure in Humans
Brief Title: Assessing Changes in Myocardial Tissue and Blood in Patients With Advanced Heart Disease
Status: Recruiting | Type: Observational
Sponsor: University of Utah (Other)
Collaborators: Intermountain Health Care, Inc. (Other); VA Salt Lake City Health Care System (U.S. Federal Agency); Hunter Holmes McGuire VA Medical Center (U.S. Federal Agency)
Responsible Party: Principal Investigator, STAVROS G DRAKOS, Principal Investigator, University of Utah
Other Study IDs: IRB_00030622
Record Dates: First submitted 2010-04-06; First posted 2010-04-08 (Estimated); Last update posted 2025-07-15 (Actual); Status verified 2025-07

CONDITIONS: Congestive Heart Failure
Keywords: Congestive Heart Failure; Left Ventricular Assist Device; LVAD; Myocardium; Remodeling; Microvasculature; Fibrosis; Cardiac Transplant
MeSH Terms: conditions — Heart Failure; Fibrosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and myocardial tissue.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Advanced Heart Failure Therapy Group: Patients diagnosed with end stage heart failure undergoing either VAD implantation or heart transplantation.
- Normal Hearts Group: Control samples will be obtained from individuals undergoing other types of cardiac surgery during which it is routine to discard some tissue intraoperatively.

SUMMARY:
Hypothesis:

Tissue and serum samples collected from end-stage heart failure patients receiving left ventricular assist device implantation (LVAD) or heart transplantation will provide information regarding the basic science of heart disease. Tissue and serum samples collected from a limited numbers of "healthy controls" (donor grafts that were not utilized for heart transplantation) will serve as a comparator in research database projects.

Design:

This is a registry project; there are no investigational treatments, drug or procedures associated with participation in registry activities. This project is an organized functional data and tissue data gathering and storing (database) endeavor with specific focus on the functional, structural, and molecular aspects of heart failure. Data collection will not immediately influence the course of treatment for any patient.

DETAILED DESCRIPTION:
Brief description of procedures:

After informed consent is obtained from the patient, the blood samples will be obtained either during a procedure from access lines inserted for the procedure or they will be drawn when other ordered lab work is done at specific time points during the study. Tissue samples will be obtained at the time of LVAD implantation by keeping the part of the left ventricular apex that the surgeon is removing in order to place the inflow cannula of the LVAD. No extra tissue sample, other than the tissue that has to be removed as a part of a standard LVAD, will be collected.

ELIGIBILITY:
Inclusion Criteria:

* >18 years of age diagnosed with heart failure undergoing either LVAD implantation or heart transplantation
* 13 to 18 years of age, specifically, older children with heart failure whose body mass index is large enough to accommodate and LVAD

Exclusion Criteria:

* Neither patient nor patient representative understands spoken English
* Neither patient nor patient's personal representative is willing to give written consent for participation.

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Either gender, ≥ 13 years of age, any ethnicity, diagnosed with end stage heart failure undergoing either VAD implantation or heart transplantation.
  Control samples will be obtained from individuals undergoing other types of cardiac sugery during which it is routine to discard some tissue intraoperatively.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2008-09 (Actual); Primary Completion 2028-01 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Change in myocardial function | baseline and 3 months
  Myocardial function, measured by left ventricular ejection fraction, will be assessed pre-LVAD implant (baseline) and compared with myocardial function assessed at 3 months post-LVAD implant

CONTACTS AND LOCATIONS:
Overall Officials: Stavros Drakos, M.D., Ph.D., Principal Investigator — University of Utah Health Sciences Center & VA Salt Lake City Health Care System
Locations (3):
- United States (3):
  - Intermountain Medical Center, Murray, Utah
  - University of Utah Health Sciences Center, Salt Lake City, Utah
  - VA Salt Lake City Health Care System, Salt Lake City, Utah

REFERENCES:
- [Derived] Gatsiou A, Tual-Chalot S, Napoli M, Ortega-Gomez A, Regen T, Badolia R, Cesarini V, Garcia-Gonzalez C, Chevre R, Ciliberti G, Silvestre-Roig C, Martini M, Hoffmann J, Hamouche R, Visker JR, Diakos N, Wietelmann A, Silvestris DA, Georgiopoulos G, Moshfegh A, Schneider A, Chen W, Guenther S, Backs J, Kwak S, Selzman CH, Stamatelopoulos K, Rose-John S, Trautwein C, Spyridopoulos I, Braun T, Waisman A, Gallo A, Drakos SG, Dimmeler S, Sperandio M, Soehnlein O, Stellos K. The RNA editor ADAR2 promotes immune cell trafficking by enhancing endothelial responses to interleukin-6 during sterile inflammation. Immunity. 2023 May 9;56(5):979-997.e11. doi: 10.1016/j.immuni.2023.03.021. Epub 2023 Apr 25. PMID 37100060